CLINICAL TRIAL: NCT06209151
Title: Procedure Related Infections in Intensive Care Unit
Brief Title: Intensive Care Unit Procedure Related Infections
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Farouk, Lecturer of critical care, Cairo University
Other Study IDs: Kasr alainy school of medicine
Record Dates: First submitted 2023-12-28; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: monitor signs of infection — Prospective observational study of 1040 patients admitted to the ICU without any signs of infection. All patients were subjected to one or more of the most used procedures in ICU (Intubation & mechanical ventilation, Central line insertion and Urinary catheterization) for at least 48 hours. Then, they were followed for any signs of infection either clinically or laboratorial.

SUMMARY:
Objectives: To identify the rate and predictors of procedure related infection, the most causative organisms and the effect on ICU stay and in hospital mortality. To show the validity of NEW score in predicting mortality.

Methods: Prospective observational study of 1040 patients admitted to the ICU without any signs of infection. All patients were subjected to one or more of the most used procedures in ICU (Intubation & mechanical ventilation, Central line insertion and Urinary catheterization) for at least 48 hours. Then, they were followed for any signs of infection either clinically or laboratorial.

DETAILED DESCRIPTION:
AIM OF THE WORK

* To identify the rate and predictors of procedure related infections in ICU after application of all preventive measures and to identify most causative organisms.
* Identification of the effect of procedure related infections on ICU stay and in hospital mortality.
* To study the validity of NEW score in predicting mortality in comparison to APACHE II score .

PATIENTS AND METHODS

Study design:

This was a prospective observational study carried out at medical and cardiac intensive care units (ICUs) of 3 secondary and tertiary care hospitals from July 2022 to June 2023 and included 1040 patients.

Inclusion criteria:

All consecutive adult patients admitted to ICU who had been subjected to the following procedures:

1. Urinary catheterization.
2. Central venous catheter (CVC) insertion.
3. Endotracheal intubation and mechanical ventilation.

Exclusion criteria:

* Patients with evidence of infection prior to ICU admission.
* Procedures done before ICU admission.

All patients were subjected to the following assessment:

A) On admission:

* The acute physiology and chronic health evaluation II (APACHE II) score.
* New early warning score 2 (NEWS2): NEWS ranges from 0, indicating the lowest severity of illness, to a maximum value of 20.
* Detailed history including age, sex, medical history.
* Complete clinical examination.
* Chest x-ray.

B) ICU stay:

• Laboratory investigations include Complete blood count (CBC), C reactive protein (CRP), renal and liver chemistry after 2, 4, 6, 12, 18 and 24 days.

Blood, urine and sputum cultures if infection was suspected.

• Chest x-ray if chest infection suspected.

C) FOLLOW UP :

* Length of mechanical ventilation
* Length of ICU stay
* Length of hospital stay
* Morbidity & mortality

Primary outcomes:

1. Identification of rate and predictors of procedure related infections.
2. Identification of the most causative organisms.

Secondary outcomes:

1. Identification of the effect of procedure related infections on ICU stay and in hospital mortality.
2. The validity of NEW score in predicting mortality

Definitions:

Ventilator associated pneumonia (VAP): was defined as pneumonia occurring >48 hours following endotracheal intubation when a new or progressive lung infiltrates, consolidation, or cavitation on chest X-ray develops in a patient with:

* New onset of purulent bronchial secretions with leukopenia (white blood cells <4×109/L) or leukocytosis (>12×109/L)
* Core temperature ≥38.5°C or ≤36°C without other cause, significant positive culture from blood, or endotracheal aspirate, broncho-alveolar lavage (BAL), or culture from another relevant site of infection [10].

Catheter associated urinary tract infection (CAUTI): A patient must meet all three criteria below:

1. Patient had an indwelling urinary catheter that had been in place for >2 days on the date of event (day of device placement=day 1) and was either present for any portion of the calendar day on the date of event or removed the day before the date of event.
2. Patient has at least one of the following signs or symptoms:

   fever (>38.0°C); suprapubic tenderness; costovertebral angle pain or tenderness; urinary urgency; urinary frequency; dysuria.
3. Patient has a urine culture with no more than two species of organisms identified, at least one of which is a bacterium of ≥105 cfu/mL.

Central line associated blood stream infection (CLABSI): A patient with a central venous catheter who has a recognized pathogen isolated from one or more blood cultures after 48 h of catheterization; or with the same skin commensals cultured from two or more blood cultures drawn on separate occasions; the pathogen is not related to an infection at another body site; and the patient has one or more of the following signs or symptoms: fever (≥38⁰c), chills, or hypotension, CLABSI was confirmed.

Statistical analysis SPSS 26.0 (SPSS Inc., an IBM Company, Chicago, IL) was used to perform the data analyses.

Baseline differences among rates were analyzed using the chi-square test for dichotomous variables and a t-test for continuous variables. 95% confidence intervals (CIs) and P values were determined for all outcomes.

Outcomes measured during the surveillance period included the incidence of overall DAIs, VAPs, CAUTIs, and CLABSIs.

DAI rates per 1,000 device-days were calculated by dividing the total number of DAIs by the total number of specific device-days and multiplying the result by 1,000 (16).

Device utilization ratios were calculated by dividing the total number of device-days by the total number of patient-days.

Device-days are the total number of days of exposure to the device (ventilator, urinary catheter, or central line) by all of the patients in the selected population during the selected time period.

Patient-days are the total number of days that patients are in an ICU during the specified time period.

Discrimination of scoring systems was assessed using the receiver operating characteristic (ROC) curve analysis for calculating the sensitivity and specificity of each score and the corresponding area under the ROC curve.

Correlations between quantitative variables were done using Spearman correlation coefficient.

Crude excess mortality of DA-HAI equals crude mortality of ICU patients with DA-HAI minus crude mortality of patients without DA-HAI.

Crude excess LOS of DA-HAI equals crude LOS of ICU patients with DA-HAI minus crude LOS of patients without DA-HAI.

Qualitative variables were presented as number and percentage (%).

ELIGIBILITY:
Inclusion Criteria:

* All consecutive adult patients admitted to ICU who had been subjected to the following procedures:

  1. Urinary catheterization.
  2. Central venous catheter (CVC) insertion.
  3. Endotracheal intubation and mechanical ventilation.

Exclusion Criteria:

* • Patients with evidence of infection prior to ICU admission.

  * Procedures done before ICU admission.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all ppopulations
Sampling Method: Non-Probability Sample
Enrollment: 1040 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Identification of rate and predictors of procedure related infections | 3 months
  1. Identification of rate and predictors of procedure related infections.
  2. Identification of the most causative organisms

SECONDARY OUTCOMES:
1. Identification of the effect of procedure related infections on ICU stay and in hospital mortality. | 3 months
  2. The validity of NEW score in predicting mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mowafy, MD, Study Director — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No